CLINICAL TRIAL: NCT01956045
Title: Critically Ill Patient's Capacity
Acronym: Capacity
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0164; 2011-A01492-39
Record Dates: First submitted 2013-07-16; First posted 2013-10-08 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Decision Making; Critical Illness
Keywords: Intensive Care Units; Judgment; Disability Evaluation; Autonomy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Decision making
  Interventions: Other: Patient's capacity

INTERVENTIONS:
Other: Patient's capacity

SUMMARY:
How to determine the decision-making capacity of critically-ill patients remain unclear. The investigator study the differences between standardised evaluation and subjective medical evaluation.

DETAILED DESCRIPTION:
After written information and consent, an independent, specially trained investigator interviews patients with a standardised test.

After written information and consent, an independent, specially trained investigator interviews residents, doctors and nurses in charge of the patient and ask them how they rates patients capacity.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers :

Doctors, hospital interns, nurses state of both sexes, aged 18 years or more working in Intensive Care, members of a social security system engaged in a clinic on the day of the assessment

* Patients :

Patients of both sexes, aged 18 years or more hospitalized in Intensive Care, members of a social security system

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically-ill patients
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
correlation between the decision-making capacity and the decision-making capacity assessed by standardized methods | at day 1
  standardized methods (patient has decision-making capacity yes/no) as described by Sessums LL, Zembrzuska H, Jackson JL. Does this patient have medical decision-making capacity? JAMA. 2011;306(4):420-427. doi:10.1001/jama.2011.1023.

SECONDARY OUTCOMES:
correlation between the global decision-making capacity evaluated by the physician in charge of the patient and the specific decision-making capacity assessed by physician in charge of the patient | at day 1
  Ability to designate a person of confidence, capacity to consent to inclusion in a research protocol, ability to participate in a discussion on the limitation therapy
association between burnout in evaluators and consistency of their decision-making capacity assessments | at day 1
Correlation between the decision-making capacity evaluated by the physician in charge of the patient, the nurse in charge of the patient and a physician not in charge of the patient | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAUTRETTE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France